CLINICAL TRIAL: NCT00296478
Title: Multi-Center, Randomized, Open-Label, Parallel Group Study of a Vaginal Micronized Progesterone Tablet (Endometrin®) Compared to Crinone 8% Vaginal Gel in Female Patients Undergoing In-Vitro Fertilization (IVF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FE999913 2004-02
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Fertility
MeSH Terms: interventions — Progesterone; Crinone

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- 1 (Experimental): Endometrin 100mg BID
  Interventions: Drug: Endometrin
- 2 (Experimental): Endometrin 100mg TID
  Interventions: Drug: Endometrin
- 3 (Active Comparator): Crinone
  Interventions: Drug: Crinone

INTERVENTIONS:
Drug: Endometrin — Endometrin 100mg BID x 10weeks
  Arms: 1
Drug: Endometrin — Endometrin 100mg TID x 10weeks
  Arms: 2
Drug: Crinone — Crinone QD x 10weeks
  Arms: 3

SUMMARY:
This multicenter, randomized, open-label study will be performed in approximately 990 healthy females undergoing IVF. Each study center will follow their study center standard practice for IVF unless otherwise noted in this protocol. The study centers will be provided with the medications for down regulation, stimulation and ovulation induction. The subjects will be randomized to study medication on the day of oocyte retrieval or the day following and will continue treatment for up to 10 weeks. The subjects with a confirmed pregnancy will be required to return to the clinic several times during the course of the 10 week treatment period for serum pregnancy tests and transvaginal ultrasounds to monitor the pregnancy.

DETAILED DESCRIPTION:
This multicenter, randomized, open-label study will be performed in approximately 990 healthy females undergoing IVF. Each study center will follow their study center standard practice for IVF unless otherwise noted in this protocol. The study centers will be provided with the medications for down regulation, stimulation and ovulation induction. The subjects will be randomized to study medication on the day of oocyte retrieval or the day following and will continue treatment for up to 10 weeks. The subjects with a confirmed pregnancy will be required to return to the clinic several times during the course of the 10 week treatment period for serum pregnancy tests and transvaginal ultrasounds to monitor the pregnancy.

ELIGIBILITY:
Inclusion Criteria

1. Pre-menopausal females between the ages of 18 and 42 years Non-smokers. For females who are past smokers, they must have stopped tobacco usage for at least 3 months prior to baseline visit.
2. Early follicular phase (day 2-4) FSH (follicle stimulating hormone) less than or equal to 15 IU/L and Estradiol within normal limits
3. LH (luteinizing hormone), PRL (prolactin), T (testosterone), DHEA-S (dehydroepiandrosterone sulfate) and TSH (thyroid-stimulating hormone), within the normal limits for the clinical laboratory, or considered not clinically significant by the investigator within 6 months prior to screening.
4. Negative serum hepatitis B surface antigen, hepatitis C antibody, HIV antibody, and rapid plasma reagin tests within 3 months prior to screening
5. Seropositive for rubella and varicella and ABO grouping and Rho (D) typing prior to screening
6. Documented history of infertility (eg, unable to conceive for at least one year or for 6 months for women ≥38 years of age or bilateral tubal occlusion or absence).
7. Male partner with recent (within 6 months prior to screening) semen analysis showing normalcy adequate for IVF by standard WHO and/or Kruger criteria. Donor sperm may be used, if indicated, provided that it meets standard WHO criteria.
8. Normal Transvaginal ultrasound at screening (or within 14 days of screening) with presence of both at least ovaries without evidence of clinically significant abnormality consistent with findings adequate for ART with respect to uterus and adnexa (no hydrosalpinx or clinically relevant uterine fibroids).
9. At least one cycle with no fertility medication prior to screening.
10. Hysterosalpingography, hysteroscopy, or sonohysterogram documenting a normal uterine cavity.
11. Negative pregnancy test on the day of pituitary down regulation (prior to administration of GnRH agonist).
12. Signed informed consent.

Exclusion Criteria

1. Requires Donor oocyte or embryo recipient; gestational or surrogate carrier
2. Undergoing blastomer biopsy and other experimental ART procedures
3. Inadequate number of oocytes defined as fewer than 3 oocytes retrieved in the study cycle
4. Presence of any clinically relevant systemic disease (eg, insulin-dependent diabetes mellitus).
5. Surgical or medical condition which in the judgment of the Investigator or Sponsor may interfere with absorption, distribution, metabolism, or excretion of the drugs to be used.
6. Subjects with a body mass index (BMI) of greater than 34 at time of Screening.
7. Previous IVF or ART failure due to related to either a sperm/fertilization problem which resulted in unsuccessful fertilization or an ART with a poor response to gonadotropins. Poor response is defined as development of less than 2 mature follicles or history of 2 previous cycle cancellations prior to oocyte retrieval due to poor response.
8. Presence of abnormal uterine bleeding of undetermined origin.
9. Current or recent substance abuse, including alcohol and tobacco. (Note: Patients who stopped tobacco usage at least 3 months prior to screening visit would be allowed).
10. History of chemotherapy (except for gestational conditions) or radiotherapy.
11. Currently breast feeding, pregnant or contraindication to pregnancy.
12. Refusal or inability to comply with the requirements of the Protocol for any reason, including scheduled clinic visits and laboratory tests.
13. For male partner, obvious leukospermia (> 2 million WBC/mL) or signs of infection in semen sample within past 2 months of pituitary down regulation; if either of these conditions exists, male should be treated with antibiotics and retested prior to his partner's pituitary down regulation.
14. Documented intolerance or allergy to any of the medications used including the study medication.
15. Participation in any experimental drug study within 60 days prior to Screening.
16. Use of any of the following medications during the pretreatment and treatment phase: hormonal drug products (use of oral contraceptives during down regulation is allowed), progesterone creams, hydrocortisone and other steroid drug products, and fertility modifiers such as insulin sensitizers.
17. History of recurrent pregnancy loss defined as 3 or more spontaneous miscarriages

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1211 (Actual)
Dates: Start 2005-07; Primary Completion 2006-04 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy. | 6 weeks

SECONDARY OUTCOMES:
Biochemical pregnancy, clinical pregnancy, pregnancy outcome. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals